CLINICAL TRIAL: NCT03831425
Title: Mitochondrial Complex I Dysfunction in Prader Willi Syndrome: A New Therapeutic Target
Brief Title: Mitochondrial Complex I Dysfunction in PWS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: unable to recruit despite multiple rounds of recruitment due to (1) not meeting inclusion/exclusion criteria (2) unwilling to participate during pandemic (3) living outside Toronto (4) involved in other PWS studies (5) no response to our messages X 3
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Foundation for Prader-Willi Research (Other)
Responsible Party: Principal Investigator, Ingrid Tein, Director, Neurometabolic Clinic, Staff Neurologist, Division of Neurology, Principal Investigator, Senior Associate Scientist, Genetics and Genome Biology Program, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1000053066
Record Dates: First submitted 2019-01-22; First posted 2019-02-05 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Prader-Willi Syndrome
Keywords: CoQ10; muscle function; attention span; quality of life
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — coenzyme Q10

STUDY DESIGN:
Intervention Model Description: prospective, randomized, double-blind, controlled, cross-over study with CoQ10 and placebo arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Sick Kids research pharmacist will be responsible for dispensing the CoQ10 capsules which will be of highest grade, purity and safety from Webber Natural Pharmaceuticals Limited. A placebo will be prepared by the Sick Kids research pharmacy and will consist of lactose-filled capsules. The CoQ10 and placebo capsules will not be identical in colour, shape or taste. However, as stated above, researchers, participants and families will be blinded to the treatment phase. They will know they are receiving one capsule for one part of the study and another capsule for the next part. No one (except the pharmacist and an unblinded study team member, who will only distribute and collect the medication given to the family (will not conduct any testing)) will know which capsule contains CoQ10 and which contains the placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coenzyme Q (Experimental): Each patient will be asked to take part in a 6 wk trial of pharmaceutical grade CoQ10 and will be randomly assigned to a start time. There will be a 6 wk washout period between treatment and placebo arms. At baseline, if this is the first arm, testing will include determination of muscle function based on our 3 min step test, muscle power (maximal jump, handgrip), strength (Queens' Square), endurance (6MWT), fatigue (PedsQL fatigue scale), physical activity level (3DPAR), attention (ADHDT scale), cognition (MoCA), physical function (CHAQ).and quality of life (PedQL). Following the 6 wk CoQ10 trial, testing will include repeat determination of all of the above as well as determination of total aerobic capacity (maximum cycle ergometry) and muscle metabolism (31P-MRS ergometry).
  Interventions: Dietary Supplement: Coenzyme Q10
- Placebo (Placebo Comparator): Each patient will be asked to take part in a 6 wk trial of placebo and will be randomly assigned to a start time. There will be a 6 wk washout period between treatment and placebo arms. At baseline, if this is the first arm, testing will include determination of muscle function based on our 3 min step test, muscle power (maximal jump, handgrip), strength (Queens' Square), endurance (6MWT), fatigue (PedsQL fatigue scale), physical activity level (3DPAR), attention (ADHDT scale), cognition (MoCA), physical function (CHAQ).and quality of life (PedQL). Following the 6 wk placebo trial, testing will include repeat determination of all of the above as well as determination of total aerobic capacity (maximum cycle ergometry) and muscle metabolism (31P-MRS ergometry).
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — 6 week trial of either treatment with CoenzymeQ.
  Arms: Coenzyme Q
Other: Placebo — 6 week trial of either treatment with Placebo
  Arms: Placebo

SUMMARY:
Prader-Willi Syndrome (PWS) is characterized by profound infantile hypotonia, growth delay, cognitive impairment, muscle weakness and exercise intolerance. Studies have suggested that a defect in energy metabolism, yet to be clarified, may be involved in its pathogenesis. Many PWS patients have received Coenzyme Q10, but the rationale for this and objective impact on cellular metabolism has not been clarified.

DETAILED DESCRIPTION:
Investigators will determine the clinical efficacy of CoQ10 in a prospective, randomized, double-blind, controlled, cross-over study. Primary outcome will include determination of muscle function based on a 3 minute step test which showed good sensitivity in the investigators' pilot study. Secondary outcomes will determine effects on muscle power (maximal vertical jump), strength (hand grip), endurance (6 Minute Walk Test), fatigue (PedsQL quality of life scale), physical activity level (3DPAR), attention (ADHDT), cognition (MOCA), and physical function (CHAQ). The investigators' subaim is to elucidate the pathophysiologic mechanisms by which clinical improvements are mediated through interrogation of underlying mitochondrial dysfunction to optimize therapies. This will include determination of total aerobic capacity (maximal graded cycle ergometry), muscle metabolic function (31P-magnetic resonance spectroscopy (MRS) of muscle to evaluate high energy phosphagen, anaerobic and aerobic exercise metabolism), mitochondrial function (serum lactate, carnitine, acylcarnitines, lactate/pyruvate ratio), and blood and urine oxidative stress markers of lipid, protein and DNA peroxidation. Investigators hypothesize that CoQ10 will lead to a clinically significant improvement in motor function, power, fatigue, habitual activity, attention span & thereby quality of life in PWS.

ELIGIBILITY:
Inclusion Criteria:

1. Consent provided
2. patients with genetically confirmed PWS aged 13 to 18 years (n=14)
3. ability to cooperate with exercise testing
4. weight > 35.0 kg
5. in good general health as evidenced by medical history
6. able to take oral medications
7. for females of reproductive potential, use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 8 weeks after the end of study intervention administration
8. for males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner during study participation and for an additional 8 weeks after the end of study intervention administration

Exclusion Criteria:

1. unable to perform exercise tests,
2. already taking CoQ10
3. having liver disease or bile duct blockage,
4. having thyroid disease or taking thyroid medications
5. presence of diabetes
6. taking antiarrhythmics or antihypertensives or anti-failure medications
7. presence of gastric disorders
8. presence of skin disorders
9. pregnancy or lactation
10. lactose intolerance
11. known allergic reaction to CoQ10 or components of preparation.
12. treatment with another investigational drug or other intervention
13. current smoker or tobacco use within 6 months
14. current cannabis user or use within 6 months
15. presence of chronic respiratory disease other than asthma
16. presence of cardiac disease with cardiac insufficiency/CHF
17. presence of MR-incompatible metal in body, metal devices or tattoos
18. presence of a bleeding disorder
19. gelatin intolerance
20. clinically significant findings in laboratory tests at screening

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Three minute step test | Baseline, week 8 (after 6 weeks on study drug or placebo), [6 week washout], week 20 (after 6 weeks study drug or placebo)
  Change in the baseline number of steps in 3 minutes of testing

SECONDARY OUTCOMES:
Vertical Jump Test | Baseline, week 8 (after 6 weeks on study drug or placebo), [6 week washout], week 20 (after 6 weeks study drug or placebo)
  Change in the baseline jumping height (centimetres)
Hand Grip Test | Baseline, week 8 (after 6 weeks on study drug or placebo), [6 week washout], week 20 (after 6 weeks study drug or placebo)
  Change in the baseline hand grip strength (kg)
6 Minute walk test | Baseline, week 8 (after 6 weeks on study drug or placebo), [6 week washout], week 20 (after 6 weeks study drug or placebo)
  Change in baseline number of metres walked in 6 minutes
Pediatric Quality of Life (PedsQL) Multidimensional Fatigue Scale | Baseline, week 8 (after 6 weeks on study drug or placebo), [6 week washout], week 20 (after 6 weeks study drug or placebo)
  Change in the baseline multi-dimensional fatigue scale; total score is reported. The higher the number, the greater the fatigue (range from 0 to 72).
Three Day Physical Activity Record (3DPAR) | Baseline, week 8 (after 6 weeks on study drug or placebo), [6 week washout], week 20 (after 6 weeks study drug or placebo)
  Change in the baseline three day recall of time (number of minutes) spent at rest, and in light, moderate and vigorous activity
SWAN Rating Scale for Attention Deficit Hyperactivity Disorder (ADHD) | Baseline, week 8 (after 6 weeks on study drug or placebo), [6 week washout], week 20 (after 6 weeks study drug or placebo)
  Change in the baseline total reported score (out of 18 items). If the sum of items 1-9 is 6 or greater, the child is likely ADHD-Inattentive type. If the sum of items 10-18 is 6 or greater, the child is likely ADHD-Hyperactive/Impulsive type. If both the sums of 1-9 and 10-18 are 6 or greater, the child is likely ADHD combined type.
Montreal Cognitive Assessment (MOCA) | Baseline, week 8 (after 6 weeks on study drug or placebo), [6 week washout], week 20 (after 6 weeks study drug or placebo)
  Change in the baseline total cognitive score out of 30 points (range 0 to 30). The higher the number, the better the cognition.
Childhood Health Assessment Questionnaire (CHAQ) | Baseline, week 8 (after 6 weeks on study drug or placebo), [6 week washout], week 20 (after 6 weeks study drug or placebo)
  Change in the baseline CHAQ score. Assessment of how an illness or condition affects child's ability to function in daily life. There are individual items in each of 8 sections (Arising, Eating, Dressing, Walking, Hygiene, Reach, Grip, Activities). Scoring of individual items ranges from 0-3 (0=from no difficulty to 3= unable to do). The higher the score, the more difficult is the task to a maximum of 3 points for each section. For each of the 8 sections, whatever the highest individual score was becomes the score of the section (max 3 points). Points are added to the section score if devices or aids are used for that section (to a maximum of 3 points). The CHAQ score is the total of the 8 sections, divided by 8 with a range from 0 points (no impact on quality of life) to 3 (large impact on quality of life) . The higher the score, the greater the impact of the illness on function.
Pediatric Quality of Life Index (PedQL) | Baseline, week 8 (after 6 weeks on study drug or placebo), [6 week washout], week 20 (after 6 weeks study drug or placebo)
  Change in baseline child quality of life using pictorial scales and comparators. The lower the score, the worse the quality of life. This is scored out of 10 cm.

OTHER OUTCOMES:
Maximal Work (measured in watts ) from incremental cycle ergometry | week 8 (after 6 weeks on study drug or placebo), [6 week washout], week 20 (after 6 weeks study drug or placebo)
  Change in the amount of work (measured in watts) in a bicycle ride to exhaustion. Participants will ride a stationary bicycle (cycle ergometer) until unable to continue. Workloads will progressively increase every minute from 'easy to pedal' to 'very hard to pedal' until participants are unable to sustain the pedalling for 1 minute. The higher the watts, the more work the participant is able to do.
31-phosphorus magnetic resonance spectroscopy (MRS) ergometry | week 8 (after 6 weeks on study drug or placebo), [6 week washout], week 20 (after 6 weeks study drug or placebo)
  Change in muscular phosphocreatine ((PCr) measured by 31P-Magnetic Resonance Spectroscopy) while performing bicycle exercise in the Magnetic Resonance scanner.
Maximal Aerobic Capacity (Oxygen Uptake (VO2) in milliliters per kilogram body weight per minute)from incremental cycle ergometry | week 8 (after 6 weeks on study drug or placebo), [6 week washout], week 20 (after 6 weeks study drug or placebo)
  Change in aerobic capacity (oxygen uptake (VO2) ml/kg/min) will be measured in a bicycle ride to exhaustion. Workloads will progressively increase every minute from 'easy to pedal' to 'very hard to pedal' until participants are unable to sustain the pedalling for 1 minute. Participants will breathe through a low resistance breathing valve and inspired and expired concentrations of oxygen and carbon dioxide will be measured to determine VO2. The higher the VO2, the higher the aerobic capacity (physical fitness).

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Tein, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No